CLINICAL TRIAL: NCT07384754
Title: Evaluation of a Novel Foot Strengthening Device for Improving Fall Risk, Balance, and Gait With Age
Brief Title: Foot Strengthening to Improve Balance and Gait in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Allison Gruber, PhD, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 26834, 23946
Record Dates: First submitted 2026-01-20; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Minimalist Footwear; Traditional Foot Exercise Program; Foot Strengthening Device (ToePro); Control Condition
Keywords: Balance; Gait; Intrinsic Foot Muscles; Minimalist footwear; Aging; Fall prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Minimalist footwear (Experimental): Participants are instructed to wear minimalist footwear during activities of daily living for 8 weeks, progressively increasing wear time according to a standardized schedule.
  Interventions: Device: Minimalist footwear
- Control (No Intervention): Participants do not receive any foot-strengthening intervention and continue usual activities.
- Foot strengthening device (ToePro) (Active Comparator): Participants use a commercially available foot-strengthening device (ToePro) for a prescribed exercise protocol over 8 weeks.
  Interventions: Device: ToePro foot strengthening device
- Foot exercise program (Experimental): Participants complete a prescribed foot and ankle strengthening exercise program targeting intrinsic and extrinsic foot muscles over an 8-week period.
  Interventions: Behavioral: Foot strengthening exercises

INTERVENTIONS:
Device: Minimalist footwear — Habitual use of low-cushion, low-structure footwear designed to increase intrinsic foot muscle engagement during daily activities.
  Arms: Minimalist footwear
Behavioral: Foot strengthening exercises — Home-based exercises including toe flexion, toe press, and arch-control movements performed several times per week.
  Arms: Foot exercise program
Device: ToePro foot strengthening device — A dense foam exercise platform designed to strengthen intrinsic foot muscles through loaded toe press exercises in lengthened muscle positions.
  Arms: Foot strengthening device (ToePro)

SUMMARY:
The goal of this clinical trial is to learn whether different foot-strengthening strategies can improve foot strength, balance, walking ability, and fall-related outcomes in middle-aged and older adults (ages 45-85 years).

The main questions it aims to answer are:

* Does foot strength change from baseline after an 8-week foot-strengthening intervention?
* Do balance, gait, and physical function improve following different foot-strengthening approaches?

Researchers will compare minimalist footwear use, a foot exercise program, a foot-strengthening device (ToePro), and no intervention to see if these interventions lead to greater improvements in foot strength, balance, gait, and fall-related outcomes than no intervention.

Participants will:

* Complete baseline and post-intervention laboratory testing of foot strength, balance, physical function, and walking gait
* Perform foot strengthening exercises or wear minimalist footwear (if applicable) five days/week for eight weeks
* Complete daily logs to record intervention compliance

DETAILED DESCRIPTION:
This randomized controlled trial evaluates the effects of multiple foot-strengthening interventions on foot strength, balance, gait, and fall-related outcomes in adults aged 45-85 years. Participants are recruited using a unified screening process and randomized to one of several intervention arms across two coordinated protocols. Interventions include habitual use of minimalist footwear, a prescribed foot exercise program, use of a commercially available foot-strengthening device (ToePro), or a no-intervention control condition.

All participants complete two in-laboratory data collection sessions conducted at baseline and after an 8-week intervention period. Laboratory assessments include measurements of foot morphology, intrinsic and extrinsic foot muscle strength, standing balance, physical function, and walking gait. Participants also complete standardized questionnaires assessing physical activity, balance confidence, fall history, and foot health. A follow-up questionnaire assessing physical activity, footwear use, foot health, and falls is administered six months after the intervention period.

During the 8-week intervention period, participants assigned to an active intervention are instructed to follow standardized intervention protocols specific to their assigned group. Physical activity levels during the intervention period are monitored for all groups using wearable activity tracking devices that record metrics such as daily step count and time spent in moderate-to-vigorous physical activity. These data are used to characterize habitual physical activity during the intervention period and to account for potential differences in overall activity levels between groups.

Intervention compliance is monitored throughout the 8-week period using self-reported compliance surveys. Participants report adherence to assigned footwear use, exercise sessions, or device use according to their intervention group. Compliance data are used to quantify adherence to the prescribed intervention protocols and to support interpretation of intervention effects.

Data from both protocols are pooled to allow direct comparison of the effects of different foot-strengthening strategies on foot strength, balance, gait, and fall-related outcomes in middle-aged and older adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults: age 45-85 years old
* Able to walk without an assistive walking device or lower limb prosthesis
* No history of foot or ankle surgery
* No history of regular minimalist footwear use
* No foot or ankle issues for which study activities may be contraindicated
* BMI <= 40

Exclusion Criteria:

* Deemed unfit for physical activity by the Physical Activity Readiness Questionnaire (PAR-Q)
* Current or history of an unresolved musculoskeletal, neurological, cardiovascular, pulmonary/respiratory, metabolic, renal condition, disease, or problem
* Use of orthotics in daily (i.e., non-athletic) footwear
* Pregnancy
* Any other disease or problems that may affect movement or the ability to exercise even at a low intensity

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Hallux Flexion Strength (Curl) | From enrollment to the end of the intervention at 8 weeks
  Change in maximal hallux (big toe) flexion strength assessed using a standardized hallux curl test (i.e., flexion at the metatarsal interphalangeal joints) with a dynamometer. Participants perform brief maximal voluntary contractions, and peak force output is recorded. Higher values indicate greater hallux curl strength.
Change From Baseline in Lesser Toes Flexion Strength (Curl) | From enrollment to the end of the intervention at 8 weeks
  Change in maximal lesser toes flexion strength assessed using a standardized lesser toes curl test (i.e., flexion at the metatarsal interphalangeal joints) with a dynamometer. Participants perform brief maximal voluntary contractions, and peak force output is recorded. Higher values indicate greater lesser toes curl strength.
Change From Baseline in Hallux Flexion Strength (Press) | From enrollment to the end of the intervention at 8 weeks
  Change in maximal hallux flexion strength assessed using a toe press test that isolates hallux flexion at the metatarsophalangeal joint. Strength is measured using a force-instrumented platform, with higher values indicating greater hallux press strength.
Change From Baseline in Lesser Toe Flexion Strength (Press) | From enrollment to the end of the intervention at 8 weeks
  Change in maximal lesser toes flexion strength assessed using a toe press test that isolates flexion at the metatarsophalangeal joints. Strength is measured using a force-instrumented platform, with higher values indicating greater lesser toes press strength.
Change From Baseline in Gait Kinetic Variables | From enrollment to the end of the intervention at 8 weeks
  Change in gait kinetic variables derived from motion capture and force measurement systems during walking. Measures include ground reaction force variables such as peak vertical force. Values reflect loading patterns during gait.
Change From Baseline in Joint Angles during Gait | From enrollment to the end of the intervention at 8 weeks
  Change in lower-limb and foot joint angles measured during walking using motion capture. Joint angles are calculated across the gait cycle and represent segmental motion of the foot and lower extremity.
Change From Baseline in Joint Range of Motion During Gait | From enrollment to the end of the intervention at 8 weeks
  Change in joint range of motion (ROM) of the foot and lower extremity measured during walking using motion capture. ROM is calculated as the difference between maximum and minimum joint angles during the gait cycle.
Change From Baseline in Stance Time During Gait | From enrollment to the end of the intervention at 8 weeks
  Change in stance time measured during walking using motion capture. Stance time represents the duration the foot remains in contact with the ground during each gait cycle.
Change From Baseline in Step Length During Gait | From enrollment to the end of the intervention at 8 weeks
  Change in step length measured during walking using motion capture. Step length is defined as the anterior-posterior distance between successive foot contacts.
Change From Baseline in Cadence During Gait | From enrollment to the end of the intervention at 8 weeks
  Change in walking cadence measured during gait analysis using motion capture. Cadence is expressed as steps per minute.
Change From Baseline in Step Width During Gait | From enrollment to the end of the intervention at 8 weeks
  Change in step width measured during walking using motion capture. Step width reflects the mediolateral distance between foot placements and is used as an indicator of gait stability.
Change From Baseline in 6-Minute Walk Test Distance | From enrollment to the end of the intervention at 8 weeks
  Change in distance walked during the 6-Minute Walk Test (6MWT), measured in meters. Greater distance indicates better functional walking capacity.
Change From Baseline in 30-Second Sit-to-Stand Test Performance | From enrollment to the end of the intervention at 8 weeks
  Change in functional lower-extremity performance assessed using the 30-Second Sit-to-Stand Test. Outcomes include the total number of completed sit-to-stand repetitions, with higher values indicating better performance.
Change From Baseline in 4-Stage Balance Test Performance | From enrollment to the end of the intervention at 8 weeks
  Change in standing balance performance assessed using the 4-Stage Balance Test. Outcomes include the ability to successfully complete progressively challenging standing positions for the required duration.
Change From Baseline in Single-Leg Heel-Raise Test Performance | From enrollment to the end of the intervention at 8 weeks
  Change in plantar flexor endurance assessed using the single-leg heel-raise test. Outcomes include the number of consecutive heel raises completed with proper form, with higher values indicating greater muscular endurance.

SECONDARY OUTCOMES:
Change From Baseline in IMU-Derived Gait Acceleration Magnitude | From enrollment to the end of the intervention at 8 weeks
  Change in gait acceleration magnitude measured using an inertial measurement unit (IMU) during walking assessments. Acceleration magnitude is derived from tri-axial accelerometer signals and reflects overall movement intensity during gait.
Footwear Minimalism (Minimalist Index) | Baseline
  Footwear minimalism assessed using the Minimalist Index (MI) rating scale applied to participants' commonly worn footwear. Higher scores indicate greater footwear minimalism.
Intervention Compliance Survey Responses | Throughout the 8-week intervention period
  Participant-reported adherence to the assigned intervention assessed using standardized, electronic compliance surveys. Survey items quantify frequency and duration of prescribed footwear use, exercise sessions, or device use during the intervention period. Higher values indicate greater adherence to the assigned intervention protocol.
FitBit-Derived Moderate-to-Vigorous Physical Activity (MVPA) | Throughout the 8-week intervention period
  Moderate-to-vigorous physical activity (MVPA) assessed using a wearable activity tracker (FitBit) during the intervention period. MVPA is quantified as minutes per day spent in moderate-to-vigorous intensity activity, summarized across the intervention period. Higher values indicate greater engagement in MVPA.
Change From Baseline in International Physical Activity Questionnaire (IPAQ) Scores | From enrollment to the end of the intervention at 8 weeks
  Change in self-reported physical activity assessed using the International Physical Activity Questionnaire (IPAQ). Outcomes include estimated time spent in physical activity at different intensity levels.
Change From Baseline in Sedentary Behavior Questionnaire (SBQ) Scores | From enrollment to the end of the intervention at 8 weeks
  Change in self-reported sedentary behavior assessed using the Sedentary Behavior Questionnaire (SBQ). Outcomes include time spent in sedentary activities across multiple daily contexts.

CONTACTS AND LOCATIONS:
Overall Officials: Allison H. Gruber, PhD, Principal Investigator — Indiana University, Bloomington
Locations (1):
- School of Public Health-Bloomington, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this time, the plan for sharing individual participant data (IPD) from this study has not been finalized. Decisions regarding IPD sharing will be informed by ongoing discussions among the study team and institutional policies. Before a specific data sharing plan can be confirmed, the study team must establish appropriate procedures to ensure participant privacy and confidentiality in accordance with institutional review board (IRB) requirements.
  Additional considerations include determining suitable methods for data de-identification, defining the scope of data and supporting documentation that could be shared, and identifying appropriate data access mechanisms that support responsible use by qualified researchers. Once these considerations have been addressed, an IPD sharing plan - including the data elements to be shared, timing of availability, and access criteria - will be finalized and made publicly available.